CLINICAL TRIAL: NCT01066559
Title: Multicentric Randomized Trial of the Impact of Hemodialysis With Polymethylmetacrylate Membrane on the Improvement of Humoral Immune Response in the Hemodialyzed Patients: Application to Hepatitis B Vaccination and Correlation to sCD40 Clearing
Brief Title: Improvement of Humoral Immune Response With Hemodialysis on BK-F Membrane: Correlation to Soluble CD40 Clearing
Acronym: HEPADIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/11
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Renal Failure; Humoral Immune Alterations
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flux polymethylmetacrylate membrane (Experimental)
  Interventions: Procedure: High flux polymethylmetacrylate membrane; Biological: Hepatitis B serological control; Biological: Seric sCD40 level
- Polysulfone membranes (Active Comparator)
  Interventions: Procedure: Polysulfone membrane; Biological: Hepatitis B serological control; Biological: Seric sCD40 level

INTERVENTIONS:
Procedure: High flux polymethylmetacrylate membrane — Patients will be hemodialysed with high flux polymethylmetacrylate membranes
  Arms: High flux polymethylmetacrylate membrane
Procedure: Polysulfone membrane — Patients be hemodialysed with polysulfone membranes
  Arms: Polysulfone membranes
Biological: Hepatitis B serological control — It will be assessed at week 16, week 20 and week 40
Biological: Seric sCD40 level — Ir will be measured at inclusion and week 12 by ELISA test according to the manufacturer instructions.

SUMMARY:
The aim of this study is to improve the humoral immune response efficiency of hemodialyzed patient by the use of PMMA membrane (BK-F) able to clear the soluble form of CD40 in a model of anti-HBV vaccination

DETAILED DESCRIPTION:
Chronic renal failure is associated with humoral immune alterations characterized by a diminished vaccine response notably against hepatitis B virus (HBV). Defects in cellular contact between immunological cells have been hypothesized to explain this observation but the precise mechanism leading to this "immunocompromised" status is not clear. The soluble form of CD40 (sCD40) is dramatically increased in the serum of uremic patients, particularly in the hemodialyzed patients. This molecule acts like an inhibitor of the CD40/CD154 contact, which is pivotal in the establishment of a proper humoral immune response. It has been shown that the most elevated sCD40 levels are associated with a lack of response to HBV vaccination in the hemodialyzed patients. The majority of the hemodialysis membranes, including high flux polysulfone membranes are unable to clear sCD40 from the sera. However, we found that the high flux polymethylmetacrylate (PMMA) membrane (BK-F Toray Medical Company, Japan) allows for sCD40 clearing.

The aim of this study is to assess the effect of dialysis on PMMA membrane on the improvement of humoral immune response through the efficiency of HBV vaccination in hemodialysed patients who were non responders to one ore more previous vaccination and its link to sCD40 clearing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, male or female
* Patient not immunized against hepatitis B despite complete well done anterior vaccination according to recommendations
* Hemodialyzed patients with hemodialysed sessions performed three times a week
* Patient able to give informed consent and affiliated to the medical insurance

Exclusion Criteria:

* Pregnant woman
* Patient never vaccinated against HBV
* Previous known hepatitis B even without anti HBs antibody (anti HBc antibody or HBs antigenemia positive)
* Active neoplasia or plasma cell dyscrasia
* VIH infection
* Known allergy to vaccine or to PMMA membrane
* Patient dialysed with PMMA membrane within three months before screening
* Necessity of acetate free biofiltration or hemodiafiltration as the technique of extrarenal epuration
* Vascular access problem with necessity of unipuncture for more than 30% of dialysis sessions.
* Patient under judicial protection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who will respond to vaccination | Week 40

SECONDARY OUTCOMES:
Percentage and the level of anti-HBs antibodies | at week 16, week 20, week 24 and week 40
Correlation between the sCD40 levels and the response to HBV vaccination | At week 12 and week 40
Correlation between albuminemia, C-Reactive Protein, lymphocytes, parathyroid hormone, chronic immunosuppressive treatment or corticoid taking and vaccinal response. | at week 12, week 24, and week 36

CONTACTS AND LOCATIONS:
Overall Officials: Valérie de PRECIGOUT, MD, Principal Investigator — University Hospital, Bordeaux, France; Pierre BORIES, MD, Principal Investigator — University Hospital, Toulouse, France; Michel RINCE, MD, Principal Investigator — University Hospital, Limoges, France; Caroline DELCLAUX, MD, Principal Investigator — Hospital, Libourne, France; Antoine POMMEREAU, MD, Principal Investigator — Clinic Saint-Augustin, Bordeaux, France; Benjamin DEROURE, MD, Principal Investigator — Clinic Delay, Bayonne, France; Hervé BONAREK, MD, Principal Investigator — Hospital, Saintes, France; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux, France
Locations (6):
- France (6):
  - CH Annonay, Annonay
  - CH de la côte Basque, Bayonne
  - CHU de Besançon, Besançon
  - Saint-Augustin Clinic, Dialyze Unit, Bordeaux
  - Pellegrin Hospital, Nephrology Unit, Bordeaux
  - Larrey Hospital, Dialyze Unit, Toulouse

REFERENCES:
- [Derived] de Precigout V, Germain C, Benard A, Lacraz A, Chauveau P, Deprele C, Seigneuric B, Pommereau A, Courivaud C, Douillet M, Taton B, Combe C, Contin-Bordes C. No Improvement of Hepatitis B Vaccination Response in Patients Dialysed with a Polymethylmethacrylate Membrane Compared to High-Flux Polysulfone: Results of the HEPADIAL Study. Blood Purif. 2020;49(3):265-271. doi: 10.1159/000504035. Epub 2019 Nov 13. PMID 31722332